CLINICAL TRIAL: NCT00864461
Title: Prevalence of Metabolic Syndrome in Down Syndrome Patients
Brief Title: Frequency of Metabolic Syndrome in Down Syndrome Patients
Status: Completed | Type: Observational
Sponsor: Universidad de Guanajuato (Other)
Responsible Party: Principal Investigator, ALEJANDRO ERNESTO MACIAS HERNANDEZ, MD, Universidad de Guanajuato
Other Study IDs: 249-08
Record Dates: First submitted 2009-03-17; First posted 2009-03-18 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Metabolic Syndrome X; Down Syndrome
Keywords: Down syndrome; Metabolic syndrome X; Insulin resistance
MeSH Terms: conditions — Metabolic Syndrome; Down Syndrome; Insulin Resistance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Case: Patients with clinical and cytogenetics diagnosis of Down syndrome, between 7 - 24 years old.
- Control: Siblings of the same gender of the case, between 7-24 years old.

SUMMARY:
The aim of this study is to assess the frequency of metabolic syndrome in Down syndrome patients because the prevalence of diabetes mellitus and obesity is higher in individuals with Down syndrome than in the general population.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Down syndrome

Exclusion Criteria:

* History of congenital cardiac defects requiring open-heart surgery
* History of gastroenterologic anomalies requiring bowel resection and/or ongoing medical intervention
* History of leukemia or other cancer
* History of hypothyroidism requiring thyroid hormone replacement

Ages: 7 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2009-09-01 (Actual); Primary Completion 2009-12-21 (Actual); Study Completion 2010-03-31 (Actual)

PRIMARY OUTCOMES:
To asses the frequency of the metabolic syndrome among Down syndrome patients. Metabolic syndrome was defined by Adult Treatment Panel III criteria modified by Halley-Castillo. | One year

SECONDARY OUTCOMES:
Evaluate the insulin resistance and insulin sensitivity using the HOMA and QUICKY methods. | One year

CONTACTS AND LOCATIONS:
Locations (1):
- School of Medicine, University of Guanajuato, León, Guanajuato, Mexico

IPD SHARING:
Plan to Share IPD: No